CLINICAL TRIAL: NCT00715312
Title: Effect of Oleic Acid on Inflammation Markers and Blood Lipid Metabolites: A Randomised, Double-Blind, Crossover Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malaysia Palm Oil Board (Other Government)
Responsible Party: Teng Kim Tiu/Ms, Malaysian Palm Oil Board (MPOB)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 625.9
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-07

CONDITIONS: Inflammation
Keywords: Inflammation; LDL; Oleic acid; Palmitic acid; trans fatty acid; C-reactive protein
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Other: Novel Olein

INTERVENTIONS:
Other: Novel Olein — A total of 70g of test oil is incorporated into cooked meal which accounts for 30-35% of calorie intake
Other: Novel Olein — A total of 70g of test oil is incorporated into cooked meal which provides 30-35% of calorie

SUMMARY:
Rationale: The effect of positional distribution of dietary fatty acids on markers of inflammation and blood lipids metabolites on diets containing fatty acids such as oleic acid that are associated with reduced risk of cardiovascular disease is not widely studied.

Hypothesis: There would be difference detected in the concentrations of markers of inflammation and blood lipid metabolites in human volunteers fed controlled diets.

Study design: A randomized, double-blind, crossover clinical trial that involves 41 healthy volunteers. The volunteers will be selected based on inclusion and exclusion criteria. They will consume controlled diets for 5 weeks that provides 15% of energy from protein, 30% of energy from fat, and 55% of energy from carbohydrates. Volunteers will be assigned to each test diets which is cooked with novel olein, palm stearin or partially hydrogenated soybean oil in random order until all three diets has consumed by each person.

Main study parameters: LDL-cholesterol

ELIGIBILITY:
Inclusion Criteria:

* Healthy and free from any disease and absence of family history for arteriosclerosis or hypertension
* Not on any medication or supplements or weight loss program
* Non smokers and alcoholics

Exclusion Criteria:

* Having some health-related problems e.g fever, flu, allergy, chronic diseases
* On some treatment or medication
* Smokers and alcoholics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
LDL-cholesterol | 5 weeks

SECONDARY OUTCOMES:
C-reactive protein | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Teng Kim Tiu, Principal Investigator — Malaysia Palm Oil Board
Locations (1):
- Malaysia Palm Oil Board, Kajang, Selangor, Malaysia